CLINICAL TRIAL: NCT02002975
Title: Actos Tablets Special Drug Use Surveillance "Metabolic Syndrome in Patients With Type 2 Diabetes Mellitus"
Brief Title: Pioglitazone Special Drug Use Surveillance "Metabolic Syndrome in Patients With Type 2 Diabetes Mellitus"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 237-016; JapicCTI-132328 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pioglitazone 15 to 30 mg: administered orally once daily before or after breakfast for 3 years.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone tablets
  Other Names: ACTOS

SUMMARY:
The purpose of this survey is to determine the onset of new cerebral and cardiovascular events and changes in metabolic syndrome parameters in patients with type 2 diabetes mellitus on long-term pioglitazone (Actos Tablets) treatment.

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of pioglitazone (Actos Tablets) in patients with type 2 diabetes mellitus, designed to determine the onset of new cerebral and cardiovascular events and changes in metabolic syndrome parameters, and to analyze the association between patient baseline characteristics, including any metabolic syndrome-related risk factors, and the onset of new cerebral and cardiovascular events in an exploratory setting.

Participants will be patients with type 2 diabetes mellitus. The planned sample size is 20000.

The usual adult dosage is 15 to 30 mg of pioglitazone administered orally once daily before or after breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have type 2 diabetes mellitus and have undergone measurements for all of the following parameters to be included in this survey:

Waist circumference, height, body weight, blood pressure, Haemoglobin A1c (HbA1c), fasting triglyceride, High-density Lipoprotein (HDL)-cholesterol

Exclusion Criteria:

* Patients meeting any of the following criteria (1) to (5) will be excluded:

  1. Patients with any contraindications to pioglitazone (Actos Tablets) treatment as specified below:

     Cardiac failure, history of cardiac failure, severe ketosis, diabetic coma or precoma, type 1 diabetes mellitus, serious hepatic dysfunction, serious renal dysfunction, severe infection, perioperative state, serious trauma, history of hypersensitivity to any ingredients of pioglitazone (Actos Tablets), pregnancy or possible pregnancy
  2. Patients aged < 20 or ≥ 75 years
  3. Patients who currently have or have had any of the following: myocardial infarction, angina pectoris, cardiomyopathy, hypertensive heart disease (including left ventricular hypertrophy with cardiac hypofunction*), atrial fibrillation, atrial flutter, valvular disease, aortic dissection, cerebral infarction, cerebral hemorrhage (including subarachnoid hemorrhage). (*Reduced cardiac function is roughly defined as having a brain natriuretic peptide [BNP] ≥ 40 pg/mL.)
  4. Patients who have taken pioglitazone (Actos Tablets) within 3 months before enrollment in this survey
  5. Patients who have been enrolled in the candesartan cilexetil (Blopress) special drug use surveillance "hypertension: survey on metabolic equivalents (MetS) (Challenge-MetS)" at each medical institution.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 18223 (Actual)
Dates: Start 2007-10-16 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1203 investigative sites in Japan, from 16 October 2007 to 30 June 2013.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus were enrolled to receive pioglitazone 15 milligram (mg) - 30 mg tablet, orally, once daily for up to 3 years.
Groups:
- Pioglitazone: Pioglitazone 15 mg - 30 mg, tablet, orally, once daily for up to 3 years before or after breakfast in participants based upon the disease severity. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Pioglitazone
Started | 18223
Completed | 17651
Not Completed | 572
Not completed — Case Report Forms Uncollected | 135
Not completed — Protocol Deviation | 437

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who had efficacy data at baseline and post-baseline (3Month) available.
Arm/Group | Pioglitazone
Number analyzed (Participants) | 17651
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7037
  Male | 10614
Region of Enrollment [Number; unit: Participants]
  Japan | 17651
Duration of Type 2 Diabetes Mellitus [Count of Participants; unit: Participants] — Mean duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported.
  Participants
    < 1 year | 3076 (17.4)
    1 - < 5 years | 5620 (31.8)
    5 - < 10 years | 3685 (20.9)
    ≥ 10 years | 2783 (15.8)
    Unknown | 2487 (14.1)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/m^2] — Body Mass Index = weight (kg)/[height (m)^2
  Kilogram (kg)/m^2 | 25.78 (4.17)
Waist Circumference [Mean (Standard Deviation); unit: Centimeter (cm)] | 89.31 (10.22)
Fasting Blood Glucose [Mean (Standard Deviation); unit: Milligram (mg)/dL] | 151.5 (47.9)
Haemoglobin A1c (HbA1c) [National Glycohemoglobin Standardization Program (NGSP)] [Mean (Standard Deviation); unit: Percent] | 8.12 (1.58)
Clinical Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 134.4 (16.0)
Clinical Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 78.5 (10.7)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 208.0 (40.6)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 54.0 (15.2)
Fasting Triglyceride [Mean (Standard Deviation); unit: mg/dL] | 157.4 (104.1)
Number of Participants Who Was Current Smoker [Count of Participants; unit: Participants] | 4041
Number of Participants Who Was Current Drinker [Count of Participants; unit: Participants] | 7112
Number of Participants Who Had Medical History or Medical Complications [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Complications defined as a disease or a health condition for each participant at the start of study. Medical history/Complications was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history/complications included all medical history/complications except for those mentioned above.
  Participants | 15051

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Met at Least One New Cerebral and Cardiovascular Events
Description: Cerebral and cardiovascular events (Macroangiopathy) include the following: Sudden death, Cerebral infarction, Cerebral hemorrhage, Subarachnoid hemorrhage, Acute myocardial infarction, Angina pectoris requiring intervention or hospitalization for treatment, Cardiac failure requiring hospitalization for treatment, Atrial fibrillation, Aortic dissection. Reported data was frequency of participants who met at least one new cerebral and cardiovascular event throughout this study.
Time Frame: From Baseline, Up to 3 Years
Population: Full Analysis Set included all participants who had efficacy data at baseline and post-baseline (3 Month) available.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 17651
Percentage of Participants | 1.01

2. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (Body Weight) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in body weight as a one of metabolic syndrome parameters and for each gender (male/female).
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: Full Analysis Set included all participants who had efficacy data at baseline and post-baseline (3 Month) available.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Pioglitazone
Number analyzed (Participants) | 13653
kg
  Male Participants: number analyzed (Participants) | 8238
  Male Participants | 1.27 (4.76)
  Female Participants: number analyzed (Participants) | 5415
  Female Participants | 1.53 (4.61)

3. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (Waist Circumference) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in waist circumference as a one of metabolic syndrome parameters and for each gender (male/female).
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: Full Analysis Set included all participants who had efficacy data at baseline and post-baseline (3 Month) available.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pioglitazone
Number analyzed (Participants) | 11418
cm
  Male Participants: number analyzed (Participants) | 6868
  Male Participants | 0.51 (5.18)
  Female Participants: number analyzed (Participants) | 4550
  Female Participants | 0.54 (6.06)

4. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (Haemoglobin A1c (HbA1c) [National Glycohemoglobin Standardization Program (NGSP)]) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in HbA1c (NGSP) as a one of metabolic syndrome parameters.
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: Full Analysis Set included all participants who had efficacy data at baseline and post-baseline (3 Month) available. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Pioglitazone
Number analyzed (Participants) | 16558
Percent | -1.04 (1.46)

5. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (Fasting Blood Glucose) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in fasting blood glucose as a one of metabolic syndrome parameters.
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 8464
mg/dL | -25.4 (48.3)

6. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (Fasting Blood Insulin Level) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in fasting blood insulin level as a one of metabolic syndrome parameters.
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micro unit/mL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1379
micro unit/mL | -1.58 (8.38)

7. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (Total Cholesterol Level) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in total cholesterol level as a one of metabolic syndrome parameters.
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 10034
mg/dL | -9.0 (39.3)

8. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (High-density Lipoprotein (HDL) Cholesterol Level) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in HDL cholesterol level as a one of metabolic syndrome parameters.
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 15679
mg/dL | 3.1 (12.0)

9. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (Fasting Triglyceride Level) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in fasting triglyceride level as a one of metabolic syndrome parameters.
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 10808
mg/dL | -28.7 (88.8)

10. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (Systolic Blood Pressure) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in systolic blood pressure as a one of metabolic syndrome parameters.
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pioglitazone
Number analyzed (Participants) | 16583
mmHg | -3.1 (16.2)

11. Primary Outcome: Changes From Baseline in Metabolic Syndrome Parameters (Diastolic Blood Pressure) at Final Assessment Point
Description: Changes from baseline in metabolic syndrome parameters at final assessment point (up to 3 years) were reported. The reported data on this outcome measure is in diastolic blood pressure as a one of metabolic syndrome parameters.
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pioglitazone
Number analyzed (Participants) | 16583
mmHg | -2.8 (10.8)

12. Secondary Outcome: Changes From Baseline in HbA1c (NGSP) With Number of Metabolic Syndrome-related Risk Factor (MetS-related Factor) at Final Assessment Point
Description: Changes from baseline in HbA1c (NGSP) with number of MetS-related factor were reported instead. Risk factors included Glucose Intolerance, Complication of Hypertension, Complication of Hyperlipidemia, Obesity, and Family History of Diabetes in Second-Degree Relatives.
Time Frame: From Baseline and final assessment point (Up to 3 Years)
Population: Full Analysis Set included all participants who had efficacy data at baseline and post-baseline (3 Month) available.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Pioglitazone
Number analyzed (Participants) | 17651
Percent
  One Factor: number analyzed (Participants) | 668
  One Factor | -0.89 (1.68)
  Two Factor: number analyzed (Participants) | 2740
  Two Factor | -1.00 (1.53)
  Three Factor: number analyzed (Participants) | 5524
  Three Factor | -1.04 (1.42)
  Four Factor: number analyzed (Participants) | 5731
  Four Factor | -1.04 (1.39)

13. Secondary Outcome: Association Between Patient Baseline Characteristics, Including Any Metabolic Syndrome-related Risk Factors, and Onset of New Cerebral and Cardiovascular Events
Time Frame: 3 Years
Population: Outcome measure, "Association between patient baseline characteristics, including any metabolic syndrome-related risk factors, and onset of new cerebral and cardiovascular events", on protocol section could not be summarized because study protocol was not defined what is the specific data for association precisely and there were no data to report.
Arm/Group | Pioglitazone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 Years
Description: Only adverse drug reactions (ADRs) were collected in this study. ADRs are adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms/diseases temporally associated with the use of a medicinal product reported throughout the study.
Arm/Group | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 82/17651
Other Adverse Events (participants affected / at risk) | 467/17651
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=17651)
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 9
Spinocerebellar disorder (Nervous system disorders) | 1
Diabetic retinopathy (Eye disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 11
Angina pectoris (Cardiac disorders) | 5
Atrial fibrillation (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 17
Cardiac failure congestive (Cardiac disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 3
Death (General disorders) | 1 — Additional Description: The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Oedema peripheral (General disorders) | 1
Sudden death (General disorders) | 7 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood calcium increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Blood potassium increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Protein urine present (Investigations) | 1
Brain natriuretic peptide increased (Investigations) | 2
Brain natriuretic peptide abnormal (Investigations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Peripheral revascularisation (Surgical and medical procedures) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=17651)
Oedema (General disorders) | 279
Oedema peripheral (General disorders) | 188

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.